CLINICAL TRIAL: NCT00878046
Title: A Non-comparative, Multi-centre Study to Evaluate the Safety and Efficacy of the DePuy Silent™ Hip Prosthesis in Primary Total Hip Replacement
Brief Title: Multi-centre Study to Assess Long-term Safety and Efficacy of the Silent™ Hip Prosthesis in Primary THR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Silent Hip has been rationalized for business reasons only
Sponsor: DePuy International (Industry)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT05/01
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis
Keywords: Hip; Cementless; Conservative
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DePuy Silent™ Hip femoral prosthesis (Experimental): A short cementless, femoral component for use in total hip arthroplasty
  Interventions: Device: DePuy Silent™ Hip femoral prosthesis

INTERVENTIONS:
Device: DePuy Silent™ Hip femoral prosthesis — A short cementless, femoral component for use in total hip arthroplasty

SUMMARY:
The purpose of this study is to determine if the Silent™ hip is effective in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments. A subset of patients will undergo scans to allow the bone mineral density of the bone surrounding the implant to be monitored

DETAILED DESCRIPTION:
The purpose of this study is to determine if the Silent™ hip, when used as part of an artificial hip joint, is effective in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments. A subset of patients will undergo scans to allow the bone mineral density of the bone surrounding the implant to be monitored

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 18 years or above at the point of screening for participation.
* Subjects who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
* Subjects who, in the opinion of the Clinical Investigator, are able to understand this clinical investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-treatment follow-ups.
* Subjects with non-inflammatory osteoarthritis of the hip who require a primary total hip replacement and are considered suitable for a cementless femoral and acetabular component.

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.
* Women who are pregnant.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical study with an investigational product in the last 6 months. This exclusion does not apply to those subjects who are participating in the pilot investigation of the DePuy Silent Hip (CT01/27)
* Subjects who are currently involved in any injury litigation claims.
* Subjects who have osteonecrosis of the femoral neck
* Subjects with significant bone loss or gross deformity in the region of the neck of the femur as identified on the pre-operative radiographs, where in the Investigator's opinion, there could be considerable migration of the DePuy Silent Hip or a significant chance of fracture of the femoral shaft and/or the lack of adequate bone to support the DePuy Silent Hip.
* Subjects with a Charnley C classification.
* Subjects with an active local or systemic infection.
* Subjects with loss of musculature, neuromuscular compromise or vascular deficiency in the affected limb rendering the arthroplasty procedure unjustified.
* Subjects with Paget's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2005-05; Primary Completion 2009-03 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Incidence of complications | 6mths post-surgery
Harris Hip score change at 6mths post-surgery | 6mths post-surgery

SECONDARY OUTCOMES:
Harris Hip Score | 3mths, 6mths, 1yr, 2yrs, 5yrs, 10yrs and 15yrs post-surgery
Oxford Hip Score | 3mths, 6mths, 1yr, 2yrs, 5yrs, 10yrs and 15yrs post-surgery
UCLA Activity Rating | 3mths, 6mths, 1yr, 2yrs, 5yrs, 10yrs and 15yrs post-surgery
Incidence of post operative radiological signs | 7 days, 3mths, 6mths, 1yr, 2yrs, 5yrs, 10yrs and 15yrs post-surgery
Change in bone mineral density | 7days, 3mths, 6mths, 1yr and 2yrs post-surgery
Kaplan-Meier Survivorship Calculations | 3 months, 6 months, and Annually

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (3):
  - Royal Newcastle Hospital, Broadmeadow
  - Prince of Wales Private Hospital, Sydney
  - Sydney Adventist Hospital, Sydney
- Hôpital Raymond Poincaré, Garches, France
- Orthopädishe Universitätsklinik, Frankfurt, Germany
- Ospedali Riuniti di Jesi, Iesi, Italy
- Llandough Hospital, Cardiff, United Kingdom